CLINICAL TRIAL: NCT05246579
Title: Prospective Evaluation of Pathways for Preterm Birth: The PEPP Study
Brief Title: Prospective Evaluation of Pathways for Preterm Birth
Acronym: PEPP
Status: Recruiting | Type: Observational
Sponsor: John O'Brien, MD (Other)
Responsible Party: Sponsor-Investigator, John O'Brien, MD, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 73519
Record Dates: First submitted 2022-01-31; First posted 2022-02-18 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Preterm Birth; Cervix; Pregnancy
Keywords: Cervical Length; Preterm Birth; Inflammation
MeSH Terms: conditions — Premature Birth; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Patients with short cervix: Patients with a short cervix identified on transvaginal ultrasound <30 mm
- Patients with a history of spontaneous preterm birth: Patients with a history of spontaneous preterm birth (<34 weeks)
- Patients with symptoms of preterm birth: Patients with preterm premature rupture of membranes or </=2 cm dilated before 34 weeks gestation.
- Control/Nulliparous: Nulliparous patients

SUMMARY:
This is a single center, prospective cohort study of pregnant patients at high risk for spontaneous preterm birth: patient's with history of spontaneous preterm birth, patient's with a short cervix and patient's symptomatic for preterm birth will be included. A control cohort of nulliparous patients without a short cervix will be recruited to provide baseline data. Plan to enroll 240 patients identified through our ultrasound unit with goal of 60 patients in each group.

DETAILED DESCRIPTION:
Patients will be approached for potential enrollment at the time of their anatomy ultrasound 18+0 and 23+6 weeks' gestation pending their obstetric history or if a transabdominal ultrasound evaluation or past transvaginal examination suggests the cervical length is less than 30 mm. Exclusion criteria will be reviewed and if none are present and the patient is considered a candidate for enrollment, informed consent will be performed. A 10-ml serum sample obtained. Before the transvaginal ultrasound, the patient will be asked to undergo a cervical washing of 3 cc of normal saline to obtain inflammatory cells followed by placement of a swab into the posterior fornix for 30 seconds. Patients who are found to have a short cervix will be prescribed standard of care medication (progesterone). Standard practice at our institution is to perform a cervical cerclage for women with a history of spontaneous preterm birth and a cervical length of =25mm at 16+0-23+6 weeks' gestation and this intervention will be continued regardless of enrollment. In addition, it is our standard to perform a cervical cerclage in women with progressive cervical change reaching a cervical length of <10 mm prior to 24+0 weeks regardless of obstetrical history. These standard practices will continue regardless of study participation.

Follow-Up Testing Visits. Additional study interventions will be collection of biomarker specimens and biophysical data. At 28 and 34 weeks gestation, the patient will undergo repeat TVU and 10-ml serum sample collection. A CRF will record the cervical length and the sonographer will be blinded to any prior cervical length measurement. A different sonographer will be utilized from the immediately preceding exam. All sonographers will complete the coursework for assessment of cervical length from either the Perinatal Quality Foundation CLEAR program or the Fetal Medicine Foundation.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age from 18 to 45 years of age.
* Singleton gestation.

Exclusion Criteria:

* Treatment with vaginal progesterone or intramuscular progestogen within the previous 4 weeks.
* History of congestive heart failure, chronic renal failure, or uncontrolled diabetes mellitus, or diabetes mellitus with evidence of end organ dysfunction secondary to vascular disease.
* Current pregnancy with a major fetal anomaly or known chromosomal abnormality.
* The subject has a marked uterine anatomic malformation that may alter pregnancy duration such as a septated uterus, unicornuate uterus, or uterine didelphys.
* The subject is considered not capable or unwilling to undergo study procedures and requirements.
* The subject is symptomatic with vaginal bleeding at enrollment visit.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Subpopulation 1: Asymptomatic women with or without a history of spontaneous preterm birth who undergo screening for preterm birth with transvaginal sonography between 18-24 weeks of gestation with a cervical length =5mm and up to and including 30mm will be eligible for enrollment.
  * Subpopulation 2: Asymptomatic with a history of early spontaneous (PTL or PROM as etiology) occurring in a prior pregnancy at 20-34 weeks' gestation.
  * Subpopulation 3: Patients with symptoms of preterm birth: preterm contractions or preterm premature rupture of membranes at less than 34 weeks.
  * Control Subpopulation: Nulliparous women with a cervical length of >30 mm
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Cytokine Profile | 18-24 weeks gestation
  Serum and Cervicovaginal cytokine profile (CRP, ICAM-1, IL-1α, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-8 (HA), IL-10, MCP-1, PIGF, TNFα, TNFβ)
Inflammatory Cytokine Profile | 28 weeks gestation
  Serum and Cervicovaginal cytokine profile (CRP, ICAM-1, IL-1α, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-8 (HA), IL-10, MCP-1, PIGF, TNFα, TNFβ)
Inflammatory Cytokine Profile | 34 weeks gestation
  Serum and Cervicovaginal cytokine profile (CRP, ICAM-1, IL-1α, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-8 (HA), IL-10, MCP-1, PIGF, TNFα, TNFβ)

SECONDARY OUTCOMES:
Progesterone Cytokine Response | 18-24 weeks gestation
  Serum and cervicovaginal cytokine profiles of those patients receiving progesterone for short cervix before and after exposure. (CRP, ICAM-1, IL-1α, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-8 (HA), IL-10, MCP-1, PIGF, TNFα, TNFβ)
Progesterone Cytokine Response | 28 weeks gestation
  Serum and cervicovaginal cytokine profiles of those patients receiving progesterone for short cervix before and after exposure. (CRP, ICAM-1, IL-1α, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-8 (HA), IL-10, MCP-1, PIGF, TNFα, TNFβ)
Progesterone Cytokine Response | 34 weeks gestation
  Serum and cervicovaginal cytokine profiles of those patients receiving progesterone for short cervix before and after exposure. (CRP, ICAM-1, IL-1α, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-8 (HA), IL-10, MCP-1, PIGF, TNFα, TNFβ)

CONTACTS AND LOCATIONS:
Overall Officials: John O'Brien, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No